CLINICAL TRIAL: NCT06968195
Title: A Phase I Clinical Trial Investigating Autologous CAR T Cells Targeting GPC3 in Relapsed or Refractory Hepatocellular Carcinoma
Brief Title: Autologous CAR T Cells Targeting GPC3 (RPCAR01) for the Treatment of Advanced or Metastatic GPC3 Expressing Hepatocellular Carcinoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: awaiting agreement with Sponsor
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3831524; NCI-2025-03008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3831524 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Recurrent Hepatocellular Carcinoma; Refractory Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Specimen Handling; Cyclophosphamide; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (RPCAR01 CAR T cells) (Experimental): Patients undergo leukapheresis within 28 days prior to RPCAR01 CAR T cell infusion. Patients then receive cyclophosphamide IV over 2 hours and fludarabine IV over 30 minutes on days -5, -4, and -3 and RPCAR01 CAR T cells IV over 15 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA during screening and blood sample collection and CT or MRI throughout the trial. Patients may also optionally undergo tissue sample collection throughout the trial.
  Interventions: Biological: Anti-GPC3-CAR Autologous T Lymphocytes; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Biological: Anti-GPC3-CAR Autologous T Lymphocytes — Given IV
  Other Names: Anti-GPC3 CAR Autologous T Cells; CAR-GPC3 T Cells; Glypican-3-specific CAR T Cells; GPC3-targeted CAR Autologous T Cells
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This phase I trial studies the side effects and best dose of RPCAR01 chimeric antigen receptor (CAR) T cells and to see how well it works in treating patients with GPC3 expressing hepatocellular carcinoma (HCC) that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). In GPC3 expressing HCC cancerous cell tissue overexpresses, or makes too much of, a protein called "GPC3" on the surface of those cells (while only rarely expressed in healthy tissue). RPCAR01 is a genetically modified T cell (a part of the immune system) product that targets GPC3 and decreases the inhibition of T cells by a protein called transforming growth factor beta (TGFB). The drug is prepared by taking T cells from the blood by a procedure called "leukapheresis." The T cells are then modified to make them target GPC3 and disrupt TGFB which may help the body's immune system identify and kill GPC3 tumor cells. Lymphodepletion chemotherapy with cyclophosphamide and fludarabine involves receiving a short course of chemotherapy to kill T cells before receiving the RPCAR01 CAR T cell infusion. Giving RCAR01 CAR T cells may be safe, tolerable, and/or effective in treating patients with advanced or metastatic GPC3 expressing HCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety, toxicity, maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of autologous genetically modified CAR T cells administered as a single infusion targeting GPC3 in adult patients with advanced or metastatic GPC3 expressing hepatocellular carcinoma.

SECONDARY OBJECTIVE:

* To assess anti-tumor activity and in vivo persistence of adoptively transferred CAR T cells.
* Safety and treatment tolerability

EXPLORATORY OBJECTIVES:

I. To assess serial serum cytokine levels and C-reactive protein (CRP) levels following CAR T cell infusions.

II. To identify biomarkers associated with treatment response. III. To investigate the milieu of the tumor microenvironment pre and post exposure to CAR T cell therapy.

IV. To assess circulating tumor-derived deoxyribonucleic acid (Ct DNA) levels pre and post CAR T cell therapy.

V. To assess circulating CAR T cell expansion and persistence.

OUTLINE: This is a dose escalation study of anti-GPC3-CAR autologous T lymphocytes (RPCAR01) CAR T cell.

Patients undergo leukapheresis within 28 days prior to RPCAR01 CAR T cell infusion. Patients then receive cyclophosphamide intravenously (IV) over 2 hours and fludarabine IV over 30 minutes on days -5, -4, and -3 and RPCAR01 CAR T cells IV over 15 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition (MUGA) during screening and blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial. Patients may also optionally undergo tissue sample collection throughout the trial.

After completion of study treatment, patients are followed up at days 2, 3, 4, 5, 6, 7, 14, and 28, months 2, 4, 6, 8, 10, and 12, and then as per separate long term follow up study for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Pathologically confirmed diagnosis of hepatocellular carcinoma. Mixed hepatocellular cholangiocarcinoma histology will be excluded in this trial
* Must have received at least 2 recommended standard of care lines of therapy for HCC which include checkpoint inhibition and a tyrosine kinase inhibitor such as lenvatinib
* Tissue confirmation of expression of GPC3 with immunohistochemistry (IHC) on archival tissue. ≥ 50% of tumor cells should be IHC 1+ or greater GPC3 intensity
* Presence of measurable disease, with Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at the time of intervention consent. Previously treated lesions are acceptable as long as there is a new confirmed measurable component
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1
* Life expectancy of at least 3 months
* Patients with chronic hepatitis B virus (HBV) infection with active disease who meet the criteria for anti HBV therapy should be on a suppressive antiviral therapy prior to initiation of therapy
* Patients with a history of hepatitis C virus (HCV) infection should have completed curative antiviral treatment and have a HCV viral load below the limit of quantification
* Patients with HIV should have CD4+ T-cell (CD4+) counts ≥ 350 cells/µL within 3 months of study enrollment
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 65,000/mcL
* Total bilirubin ≤ 1.5 x 1.3 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional upper limit of normal (ULN)
* Creatinine clearance ≥ 50 mL/min (Cockroft-Gault)
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients eligible for curative surgical or locoregional treatment options at the time of screening will not be included in the clinical trial.
* Patients with underlying Child-Pugh B or C liver cirrhosis (score of 7 or over)
* Patient does not have archival tumor tissue available for GPC3 testing
* Patients with a recent history of ongoing active bleeding
* Patients who have a current medical history of alcohol abuse
* Patient with a history of grade 2 or greater immune mediated toxicities of a major organ or a history of autoimmune hepatitis, pneumonitis or myocarditis
* Participants who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. A washout period of 2 weeks is required prior to leukapheresis
* Participants with known leptomeningeal disease or brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Concomitant systemic glucocorticoid use at a dose equivalent to > 10 mg daily prednisone at the time of leukapheresis and/or within 4 weeks of CAR T infusion
* Clinical or radiographic evidence of bowel obstruction or need for parenteral hydration and/or nutrition
* Active autoimmune disease
* Prior history of seizure disorder
* Pregnancy or breast-feeding female participants
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of anti-GPC3 targeted chimeric antigen receptor (CAR) T cells | Up to 30 days following T cell infusion
  Will be determined based on the treatment-emergent toxicity (defined by Common Terminology Criteria for Adverse Events [CTCAE] version 5) occurring during the 30-day period following the initial T cell infusion.
Recommended phase 2 dose (RP2D) | Up to 30 days following T cell infusion
  MTD and secondary endpoints will inform selection of RP2D. The MTD is defined as the highest dose with an observed incidence of dose limiting toxicity (DLT) in no more than one out of six patients treated at a particular dose level. The MTD will be identified using the standard 3+3 design.
DLT | Up to 30 days following T cell infusion
  DLTs will be summarized by dose level using frequencies and relative frequencies.
Incidence of adverse events | Up to 1 year following T cell infusion
  All patients who received any dose of anti-GPC3 CAR T cells infusion will be considered evaluable for safety analysis. CTCAE will be utilized for adverse event reporting. All adverse events will be summarized by dose levels, attribution, and grade using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Objective response rate | Up to 15 years
  As determined by Response Evaluation Criteria in Solid Tumors and Immune-Modified Response Evaluation Criteria in Solid Tumors. Will be summarized overall and by dose level using frequencies and relative frequencies using simple relative frequencies. The corresponding 95% confidence intervals for the estimated probabilities will be computed using the Clopper-Pearson method.
Overall survival | From treatment initiation until death due to any cause or last follow-up, assessed up to 15 years
  Will be summarized in the overall sample and by dose level using standard Kaplan-Meier curves.
Progression-free survival | From treatment initiation until disease progression, death, or last follow-up, assessed up to 15 years
  Will be summarized in the overall sample and by dose level using standard Kaplan-Meier curves.
Percentage of patients with detectable versus (vs.) undetectable anti-GPC3 CAR T cells | At days 2, 4, 7, and 14, months 2 and 6, and 1 year
  To assess the in vivo persistence of anti-GPC3 CAR T cells, the percentage of patients with detectable vs. undetectable anti-GPC3 CAR T cells at each time point will be evaluated in the efficacy analysis set. The abundance of anti-GPC3 CAR T cells will be analyzed at each time point. Summary statistics and graphical measures will be used to describe the T-cell persistence, T cell differentiation, memory, and exhaustion over time. Will be summarized overall and by dose levels using mean and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Krishnamurthy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States